CLINICAL TRIAL: NCT01929785
Title: Application of In-House Developed Nanomedicine Technology for Diagnosis and Management of Post-Transplant Heart Allograft Patients
Brief Title: BIIR Gene to Manage Heart Allograft Patients
Status: Completed | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 009-265
Record Dates: First submitted 2013-01-31; First posted 2013-08-28 (Estimated); Last update posted 2016-01-13 (Estimated); Status verified 2016-01

CONDITIONS: Cardiac Transplant Failure
Keywords: post tranplant heart allograft

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — To create new means to detect rejection at the earliest stages, to help prevent progression through earlier treatment, to discover new avenues targets for treatment of heart graft rejection, and to reduce the cost of post-transplant health care
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Pre and Post Transplant: Research blood samples will be drawn pre-transplant, and at monthly post transplant visits at times corresponding to post-transplant, standard of care ImmKnowo and AlloMap clinical testing. A minimum of 12 visits per patient is expected
- One year post transplant: The second group will include heart transplant recipients at one year post transplant who consent to participate in the study. Research blood samples will be drawn at quarterly post transplant visits (standard of care in Year 2 post transplant) corresponding to ImmunKnow and AlloMap testing. A minimum of 4 visits per patient is expected.

SUMMARY:
This is a single center observational study. Duration of the study is 1 year. Participants will be followed in 2 groups. Group 1 will include all patients who have undergone a heart transplant, through the first year post transplant. Group 2 will include heart transplant recipients from 1 year to 2 years post transplant. Groups will be enrolled simultaneously. It is anticipated each group will have 25 participants.

DETAILED DESCRIPTION:
Application of the BIIR gene expression profile approach to heart transplantation clinical diagnostic issues is likely to create new means to detect rejection at the earliest stages, to help prevent progression through earlier treatment, to discover new avenues targets for treatment of heart graft rejection, and to reduce the cost of post-transplant health care

ELIGIBILITY:
Inclusion Criteria:

* Patients who will have or have already received a heart transplant.
* Patients who have no other transplant history.
* Men and Women ages 18 to 73

Exclusion Criteria:

* Patients who are pregnant or lactating will not be eligible for this protocol.
* Patients who are cognitively impaired

Ages: 18 Years to 73 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heart transplant patients from Baylor University Medical Center,Dallas
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2009-12; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
To systematically collect blood samples from heart allograft recipients who are 0-2 years post-transplant to create a repository for genomic research. | 2 years
  To systematically collect blood samples from heart allograft recipients who are 0 -2 years post-transplant for eventual screening of blood cell gene activity, in order to identify diagnostically useful biomarkers that can help distinguish among multiple possible clinical presentation, e.g., acute rejection, antibody mediated rejection, infection, coronary artery disease, a variety of potential causes for heart dysfunction.).

SECONDARY OUTCOMES:
Recent work using our gene expression profiling (GEP) has shown that peripheral blood cells display a unique GEP that is 90% accurate for detection of acute rejection in liver transplant patients & hopefully hearts as well. | 2 years
  Recent work using our gene expression profiling (GEP) has shown that peripheral blood cells display a unique GEP that is 90% accurate for detection of acute rejection in liver transplant patients. The Investigators hypothesize that heart allograft recipients will display a similar pattern (Aim #2). The Investigators will retrospectively select longitudinal samples collected in Aim #1 from patients who did not experience rejection and from those who did, in order to determine if their GEP correlates with what we have observed for liver patients.

OTHER OUTCOMES:
To correlate the BUMC GEP results with AlloMap results. | 2 years
  To correlate the BUMC GEP results with with AlloMap results. The Investigators will retrospectively select longitudinal samples collected in Aim #1 from patients who had normal vs. high AlloMap scores
To determine whether immune response status, as reflected by donor specific antibody response adn Cylex ImmuKnow assay, alters the GEP in heart transplant patients. | 2 years
  To determine whether immune response status, as reflected by donor specific antibody response and Cylex ImmuKnow assay, alters the GEP heart transplant patients.

CONTACTS AND LOCATIONS:
Overall Officials: Shelley Hall, MD, Study Chair — Baylor Health Care System
Locations (1):
- Baylor University Medical Center, Dallas, Texas, United States